CLINICAL TRIAL: NCT07290023
Title: Characterization of the Oral and Gut Microbiota in Individuals With Serrated Polyposis Syndrome.
Brief Title: Oral and Gut Microbiota in Individuals With Serrated Polyposis Syndrome.
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)400/2020
Record Dates: First submitted 2025-12-04; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer; Serrated Polyposis Syndrome; Intestinal Microbiota
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Biological samples from saliva, and feces will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Serrated polyposis syndrome: Clinical, histological, and endoscopic data will be recorded, and biological samples from saliva, and feces will be collected.
- Individuals with sporadic serrated lesions: Clinical, histological, and endoscopic data will be recorded, and biological samples from saliva, and feces will be collected.
- Individuals with adenomas: Clinical, histological, and endoscopic data will be recorded, and biological samples from saliva, and feces will be collected.
- Individuals without polyps: Clinical and endoscopic data will be recorded, and biological samples from saliva, and feces will be collected.

SUMMARY:
* Background: Serrated polyposis syndrome is the most common colorectal polyposis syndrome. Its pathogenesis is still unknown and its diagnosis is based on clinical criteria. Despite advances in its knowledge, the intestinal microbiota of these patients has not been characterized, nor has the role of Fusobacterium nucleatum in their lesions been evaluated.
* Aim: The main objective is to compare the composition of the intestinal and oral microbiota of individuals diagnosed with serrated polyposis syndrome with individuals with sporadic serrated polyps, adenomatous polyps and without polyps. Among the secondary objective is to establish the prevalence of Fusobacterium nucleatum in oral and fecal samples.
* Methodology: Observational, case-control and multicenter study. Prospective inclusion for 24 months of all patients diagnosed with serrated polyposis syndrome, associated with three control groups: individuals without polyps, individuals with sporadic serrated lesions and individuals with adenomas. Clinical, histological, and endoscopic data will be recorded, and biological samples from saliva, and feces will be collected.

ELIGIBILITY:
Inclusion Criteria:

- Individuals who meet the diagnostic criteria for serrated polyposis syndrome and who have a recent colonoscopy (<3 months) in which at least one serrated lesion is resected (defined as hyperplastic polyp or sessile serrated lesion / polyp) proximal to the rectum ≥ 5 mm.

2) Individuals who have a recent colonoscopy (<3 months) in which it is at least dry a serrated lesion proximal to the rectum ≥ 5 mm. Must not present ≥ 5 serrated lesions metachronous or synchronous. 3) Individuals who have had a recent colonoscopy (<3 months) with resection of the less one adenoma ≥ 5 mm. 4) Individuals who have had a recent colonoscopy (<3 months) without polyps.

Exclusion Criteria:

* Suspicion of hereditary syndromes of predisposition to CRC (> 20 metachronous adenomas, Familial adenomatous polyposis, Lynch syndrome, Peutz-Jeghers syndrome, Cowden, juvenile polyposis).
* Consumption of antibiotics, probiotics or prebiotics in the last 3 months.
* Incomplete colonoscopy or with inadequate preparation in some section.
* Adenomatous, serrated or indeterminate polyps synchronous in the inclusion colonoscopy except in the group of serrated polyposis syndrome.
* Colorectal cancer or hamartomatous polyps in inclusion colonoscopy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gastroenterology consultations patients.
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Characterization of Intestinal Microbiota through 16S Sequencing | 1 year
  Characterization of Intestinal Microbiota through 16S Sequencing
Characterization of Oral Microbiota through 16S Sequencing | 1 year
  Characterization of Oral Microbiota through 16S Sequencing

SECONDARY OUTCOMES:
Quantitative Polymerase Chain Reaction (qPCR) from F. nucleatum. | 1 year
  Quantitative Polymerase Chain Reaction (qPCR) from F. nucleatum in saliva and feces.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Aguilera Castro, Principal Investigator — Vall d'Hebron Research Institute Barcelona, Spain, 08035
Locations (1):
- Lara Aguilera Castro, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cullin N, Azevedo Antunes C, Straussman R, Stein-Thoeringer CK, Elinav E. Microbiome and cancer. Cancer Cell. 2021 Oct 11;39(10):1317-1341. doi: 10.1016/j.ccell.2021.08.006. Epub 2021 Sep 9. PMID 34506740
- [Result] He X, Wu K, Ogino S, Giovannucci EL, Chan AT, Song M. Association Between Risk Factors for Colorectal Cancer and Risk of Serrated Polyps and Conventional Adenomas. Gastroenterology. 2018 Aug;155(2):355-373.e18. doi: 10.1053/j.gastro.2018.04.019. Epub 2018 Apr 24. PMID 29702117
- [Result] Avelar-Barragan J, DeDecker L, Lu ZN, Coppedge B, Karnes WE, Whiteson KL. Distinct colon mucosa microbiomes associated with tubular adenomas and serrated polyps. NPJ Biofilms Microbiomes. 2022 Aug 29;8(1):69. doi: 10.1038/s41522-022-00328-6. PMID 36038569